CLINICAL TRIAL: NCT05609123
Title: Endothelial Glycocalyx Status and Damage in Brain Death Organ Donors
Brief Title: Endothelial Glycocalyx Damage in Brain Death Organ Donors
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, David Astapenko, MD, PhD, Deputy Head for Science and Research, University Hospital Hradec Kralove
Other Study IDs: CooperatioUK_DBD_GCX
Record Dates: First submitted 2022-10-29; First posted 2022-11-08 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Brain Damage Due to Hypoxia; Organ Donors; Organ Transplant Failure or Rejection
MeSH Terms: conditions — Hypoxia, Brain; Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Brain dead organ donors: Patients with clinically proven bain death were assigned to the paraclinical confirmatory investigation of the brain death and subsequently accepted into the transplantation program.
  Interventions: Diagnostic Test: Endothelial glycocalyx damage assessment

INTERVENTIONS:
Diagnostic Test: Endothelial glycocalyx damage assessment — Degradation products of endothelial glycocalyx will be assessed in the blood and urine.

SUMMARY:
The study aims the assessment of endothelial glycocalyx (EG) degradation in deceased organ donors. There is a lack of organs for the transplantation program. By the description of the EG status, we can open room for organ optimization before transplantation and improve the organ function after transplantation in marginal donors.

ELIGIBILITY:
Inclusion Criteria:

* patients in critical condition declared as brain dead by clinical examination

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the intensive care unit with intracranial pathology are predisposed to brain death. In a time of confirmed brain death by clinical examination, the patients will be enrolled. Confirmatory paraclinical study of brain death is not mandatory for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Markers of endothelial glycocalyx damage | baseline at the time of inclusion
  Levels of syndecan-1 in serum and urine

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia